CLINICAL TRIAL: NCT03536442
Title: Examining the Impact of Trauma-informed Cognitive Behavioural Therapy Among At-risk Pregnant Women on Perinatal Mental Health Outcomes: A Pilot Study
Brief Title: Promoting Attachment Through Healing
Acronym: PATH
Status: Completed | Type: Observational
Sponsor: Western University, Canada (Other)
Collaborators: London Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Kim Jackson, Assistant Professor, Western University, Canada
Other Study IDs: 10016616; R5498A03 (Other Grant/Funding Number: Women's Xchange $15K Challenge Grant)
Record Dates: First submitted 2017-05-08; First posted 2018-05-24 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Stress Disorders, Post-Traumatic; Depressive Disorder; Anxiety Disorders
Keywords: antenatal; postpartum; mental health
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depressive Disorder; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention (CBT): As there is only one arm in this trial, this will be described in "intervention".

SUMMARY:
Intimate partner violence (IPV) is a significant and pervasive public health challenge and is associated with mental illnesses such as depression, anxiety and posttraumatic stress disorder (PTSD). Although the perinatal period may be a time of greater risk for experiencing IPV, and greater vulnerability to PTSD symptomatology, a lack of research exists pertaining to the identification/treatment of IPV-related PTSD symptoms during this period. Utilizing a mixed-methods approach, and employing a feminist, intersectional framework, the effectiveness of trauma-informed cognitive behavioural therapy (CBT) among pregnant survivors of IPV experiencing PTSD symptomatology on depression, anxiety, PTSD and maternal-infant attachment will be explored.

DETAILED DESCRIPTION:
IPV is a pervasive public health problem [1], with estimates of approximately 50% of Canadian women experiencing IPV at least once during their lifetime [2]. Some studies suggest that the perinatal period is a time of higher risk for experiencing IPV [3-4]. Numerous studies have linked women's experience of IPV with mental health concerns such as depression, anxiety and PTSD [5-8] and rates of PTSD are higher for perinatal women compared to the general population [9-10]. Prevalence rates of PTSD among survivors of IPV range from 31-84% [7,11].

The perinatal period may relate to greater risk for re-triggering of PTSD, given the physical/emotional changes, and the intimate/invasive nature of perinatal care. Additionally, the medicalized processes involved may contribute to feelings of powerlessness and vulnerability, further compromising at-risk women [9]. PTSD can alter psychological functioning and is associated with depression [12], disordered eating, substance abuse, sexual risk exposures and re-victimization [13] and failure to engage in health promotion strategies such as exercise, diet and routine health care [14]; all of which may exacerbate obstetrical risk. Furthermore, mental illness and trauma have been associated with infant prematurity, low birth weight and childhood developmental delays [15] in addition to adverse effects on maternal functioning such as maternal-child attachment [15]. As such, there are enormous personal and societal costs associated with PTSD related to IPV for childbearing women.

Recently, a significant gap in the literature was identified pertaining to the identification and treatment of IPV-related PTSD of childbearing women [16]. There is a critical need for individualized, trauma-informed care to facilitate optimal maternal and child attachment outcomes [16]. Fortunately, effective PTSD treatments exist, such as CBT; however, research exploring CBT in pregnant populations is lacking [17]. As such, the purpose of this study is to explore the effectiveness of CBT for the treatment of IPV-related PTSD among antenatal women.

ELIGIBILITY:
Inclusion Criteria:

Women who received antenatal CBT treatment from the Perinatal Nurse Specialist at the Perinatal Mental Health Clinic (London Health Sciences Centre, London, ON, Canada) who are:

* English speaking
* Have symptoms consistent with PTSD, depression, and/or anxiety

Exclusion Criteria:

* Women will be excluded if there is, or if it anticipated that there will be involvement in child protection services under the Child and Family Services Act

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — This study applies to postpartum women
Study Population: Women will be recruited from the perinatal clinic at London Health Sciences (LHSC), London, Ontario, Canada. London, Ontario is an urban setting with a population of approximately 350,000. LHSC is one of Canada's largest acute-care teaching hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
PTSD | Up to 52 weeks postpartum
  PTSD severity will be measured using the PTSD Checklist - Civilian Version

SECONDARY OUTCOMES:
Maternal-infant attachment | Up to 52 weeks postpartum
  Maternal-infant attachment will be measured using the Maternal Attachment Inventory
Presence of postpartum depression | Up to 52 weeks postpartum
  Presence of depressive symptoms will be measured using the Edinburgh Postnatal Depression Scale (EPDS). Scores greater than 12 on the EPDS will be considered positive for postpartum depression. Scores between 0-12 will be considered "low probability of depression", scores 13 and above (13-30) will be considered "high probability of depression"
Anxiety | Up to 52 weeks postpartum
  Severity of anxiety will be measured using the State-Trait Anxiety Inventory

OTHER OUTCOMES:
Maternal quality of life | Up to 52 weeks postpartum
  Maternal quality of life will be measured using the World Health Organization Quality of Life - Brief questionnaire (WHOQOL-BREF). Higher scores denote higher quality of life. We are not using a cutoff score for this measure, as it is an exploratory question and we are only looking at trends in the data, and not statistically different results among groups.
Maternal coping | Up to 52 weeks postpartum
  Maternal coping will be measured using the proactive coping inventory

CONTACTS AND LOCATIONS:
Overall Officials: Kimberley T Jackson, PhD, Principal Investigator — University of Western Ontario, Canada
Locations (1):
- London Health Sciences, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] World Health Organization. World report on violence and health. Geneva: World Health Organization; 2002
- [Background] Garcia-Moreno C, Jansen HA, Ellsberg M, Heise L, Watts CH; WHO Multi-country Study on Women's Health and Domestic Violence against Women Study Team. Prevalence of intimate partner violence: findings from the WHO multi-country study on women's health and domestic violence. Lancet. 2006 Oct 7;368(9543):1260-9. doi: 10.1016/S0140-6736(06)69523-8. PMID 17027732
- [Background] Campbell JC. Health consequences of intimate partner violence. Lancet. 2002 Apr 13;359(9314):1331-6. doi: 10.1016/S0140-6736(02)08336-8. PMID 11965295
- [Background] Afifi TO, MacMillan H, Cox BJ, Asmundson GJ, Stein MB, Sareen J. Mental health correlates of intimate partner violence in marital relationships in a nationally representative sample of males and females. J Interpers Violence. 2009 Aug;24(8):1398-417. doi: 10.1177/0886260508322192. Epub 2008 Aug 15. PMID 18718882
- [Background] Coker AL, Smith PH, Thompson MP, McKeown RE, Bethea L, Davis KE. Social support protects against the negative effects of partner violence on mental health. J Womens Health Gend Based Med. 2002 Jun;11(5):465-76. doi: 10.1089/15246090260137644. PMID 12165164
- [Background] Golding JM. Intimate partner violence as a risk factor for mental disorders: A meta-analysis. J Fam Violence. 1999;6:81-95.
- [Background] Plichta SB. Intimate partner violence and physical health consequences: policy and practice implications. J Interpers Violence. 2004 Nov;19(11):1296-323. doi: 10.1177/0886260504269685. PMID 15534333
- [Background] Seng JS, Rauch SA, Resnick H, Reed CD, King A, Low LK, McPherson M, Muzik M, Abelson J, Liberzon I. Exploring posttraumatic stress disorder symptom profile among pregnant women. J Psychosom Obstet Gynaecol. 2010 Sep;31(3):176-87. doi: 10.3109/0167482X.2010.486453. PMID 20482290
- [Background] Seng JS, Sperlich M, Low LK. Mental health, demographic, and risk behavior profiles of pregnant survivors of childhood and adult abuse. J Midwifery Womens Health. 2008 Nov-Dec;53(6):511-21. doi: 10.1016/j.jmwh.2008.04.013. PMID 18984507
- [Background] Jones L, Hughes M, Unterstaller U. Post-traumatic stress disorder (PTSD) in victims of domestic violence. Trauma, Violence, Abuse. 2001;2(2):99-119
- [Background] Breslau N, Davis GC, Peterson EL, Schultz LR. A second look at comorbidity in victims of trauma: the posttraumatic stress disorder-major depression connection. Biol Psychiatry. 2000 Nov 1;48(9):902-9. doi: 10.1016/s0006-3223(00)00933-1. PMID 11074228
- [Background] Ahluwalia IB, Merritt R, Beck LF, Rogers M. Multiple lifestyle and psychosocial risks and delivery of small for gestational age infants. Obstet Gynecol. 2001 May;97(5 Pt 1):649-56. doi: 10.1016/s0029-7844(01)01324-2. PMID 11339910
- [Background] Rheingold A, Acierno R, Resnick H. Trauma, posttraumatic stress disorder, and health risk behaviors. 2004 [cited 2016 Sep 14]; Available from: http://psycnet.apa.org/psycinfo/2003-88426-009
- [Background] Lee King PA, Duan L, Amaro H. Clinical needs of in-treatment pregnant women with co-occurring disorders: implications for primary care. Matern Child Health J. 2015 Jan;19(1):180-7. doi: 10.1007/s10995-014-1508-x. PMID 24770992
- [Background] Jackson K, Mantler T. Examining the Impact of Posttraumatic Stress Disorder Related to Intimate Partner Violence on Antenatal, Intrapartum and Postpartum Women: A Scoping Review. J Fam Violence [Internet]. 2016
- [Background] Lapp LK, Agbokou C, Peretti CS, Ferreri F. Management of post traumatic stress disorder after childbirth: a review. J Psychosom Obstet Gynaecol. 2010 Sep;31(3):113-22. doi: 10.3109/0167482X.2010.503330. PMID 20653342
- [Background] McFarlane J, Parker B, Soeken K, Bullock L. Assessing for abuse during pregnancy. Severity and frequency of injuries and associated entry into prenatal care. JAMA. 1992 Jun 17;267(23):3176-8. doi: 10.1001/jama.267.23.3176. PMID 1593739
- [Derived] Jackson KT, Parkinson S, Jackson B, Mantler T. Examining the Impact of Trauma-Informed Cognitive Behavioral Therapy on Perinatal Mental Health Outcomes Among Survivors of Intimate Partner Violence (The PATH Study): Protocol for a Feasibility Study. JMIR Res Protoc. 2018 May 25;7(5):e134. doi: 10.2196/resprot.9820. PMID 29802091